CLINICAL TRIAL: NCT04624815
Title: Factors Issued From Functional Exploration Associated to SAHOS in Asthmatic Children
Acronym: SASTHMA
Status: Terminated | Type: Observational
Why Stopped: logistics problems
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190828; IDRCB: 2019-A01976-51 (Registry Identifier: ANSM)
Record Dates: First submitted 2020-10-15; First posted 2020-11-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2020-10

CONDITIONS: Asthma; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Asthma; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
There is an increase in the prevalence of obstructive apnea-hypopnea syndrome (OSA) in children for which the pathophysiological explanation is unknown. The main objective is to compare pharyngeal collapsibility in asthmatic children with SHS score > 2.75 or ≤ 2.75 (OSA prediction score validated in French). Secondary objectives: Compare pharyngeal size, tracheal size, loop gain and its components (controller, plant), lung volumes and expired and nasal NO in asthmatic children with SHS score > 2.75 or ≤ 2.75. The bias due to the possible existence of an alveolar hyperventilation syndrome associated with asthma will be taken into account.

DETAILED DESCRIPTION:
Detailed measurements and questionnaires: Measurement of pharyngeal volume by acoustic pharyngometry in sitting and lying position with calculation of pharyngeal compliance. Measurement of ventilation (15 minutes) and transcutaneous PCO2 measurement, three apnea tests at the end of the test, hyperventilation test. PFT with spirometry and static volume measurement. Multiple flow measurement of exhaled NO with calculation of bronchial flow and alveolar fraction of NO. Nasal NO measurement. Questionnaires for OSA: the Pediatric Sleep Questionnaire (PSQ) and the SCR (Sleep Clinical Record). Questionnaires for functional respiratory disorder: French hyperventilation questionnaire SHAPE and the Nijmegen score

ELIGIBILITY:
Inclusion Criteria:

* Confirmed asthma established on the notion of typical respiratory functional signs and the notion of reversibility of a bronchial obstruction on previous PFT and/or asthma exacerbation diagnosed by the physician in an emergency room. Ongoing asthma treatment (including SABA on demand)

Exclusion Criteria:

* not asthmatic children

Ages: 6 Years to 12 Years | Sex: All
Age Groups: Child
Study Population: asthmatic children
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
pharyngeal collapsibility pharyngeal collapsibility pharyngeal collapsibility | 1 year
  Pharyngeal compliance will be measured using acoustic pharyngometry

CONTACTS AND LOCATIONS:
Overall Officials: Christophe DELCLAUX, MD-PhD, Principal Investigator — Assistance Public Hôpitaux de Paris
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No